CLINICAL TRIAL: NCT06012370
Title: A Pilot Study of Injecting Plasma-rich Platelets and Hyaluronic Acid for Patients With Stress INCONTINENCE; A NON-RANDOMIZED CLINICAL TRIAL
Brief Title: Injecting Plasma-rich Platelets & Hyaluronic Acid for Patients With Stress Urinary Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, suzy abdelaziz Abdelhamid, Assistant professor doctor, Kasr El Aini Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBH-1572023
Record Dates: First submitted 2023-08-14; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Stress Incontinence, Female
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stress incontinence patients (Other): PRP injection
  Interventions: Procedure: PRP injection

INTERVENTIONS:
Procedure: PRP injection — Injection of PRP and hyaluronic acid

SUMMARY:
Injection of PRP and hyaluronic acid in stress incontinence patients

DETAILED DESCRIPTION:
Operative details Dissection of the ant vag wall from the urethra and lower part of the bladder Identify the bladder neck using Foly s catheter injection of 1.5 to 2 ml PRP combined with Hyaluronic acid suburethra almost at the level of mid urethra (avoiding the bl neck) then closure of the vag wall ( after removal of the excess vag tissue.

ELIGIBILITY:
Inclusion Criteria:

* stress incontinence patients

Exclusion Criteria:

* prolapse patients

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Stress incontinence change | 6 months
  Visual Assessment System assessment